CLINICAL TRIAL: NCT04476485
Title: A Newly Discovered Clinical Recurrence Predictor for High-risk Hormone Receptor-positive Breast Cancer: a Real Word Study
Brief Title: Sj-subway, a Predictor for the Recurrence of High-risk Hormone Receptor-positive Breast That is Sensitive to Extended Endocrine Therapy
Status: Recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Director, Shengjing Hospital
Other Study IDs: ShengjingH 3
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
Keywords: receptor, estrogen; endocrine therapy; aromatase inhibitor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- experimental group: If the expression of sj-subway in the surgical wax block is eligible, it is recommended but not mandatory that patients follow the guidelines to choose the appropriate extended endocrine therapy.
  Interventions: Other: endocrine therapy

INTERVENTIONS:
Other: endocrine therapy — If the expression of sj-subway in the surgical wax block is eligible, it is recommended but not mandatory that patients follow the guidelines to choose the appropriate extended endocrine therapy. 1. For postmenopausal patients: Extend treatment with aromatase inhibitors 10 years: letrozole or anastrozole or exemestane. 2. For premenopausal patients: An initial 5 years tamoxifen treatment followed by additional 5 years extended tamoxifen treatment. Postmenopausals are treated with aromatase inhibitors 5 years. 3. For patients have completed ovarian function suppression plus initial 5-year aromatase inhibitor treatment: Menopausals: Aromatase inhibitors; Non-menopausals: 5 years of tamoxifen treatment or ovarian function suppression plus 5 years of aromatase inhibitor treatment. 4. For patients have completed ovarian function suppression plus initial 5-year tamoxifen treatment: Menopausals: Aromatase inhibitors for additional 5 years; Non-menopausals: Tamoxifen for additional 5 years.

SUMMARY:
Hormone receptor-positive breast cancer accounts for about 70% of all breast cancers. Extended endocrine therapy with aromatase inhibitor is the current main treatment for hormone receptor-positive breast cancer. However, previous studies have shown a long-lasting risk of the recurrence of hormone receptor-positive breast cancer at early stage, and disease recurrence is considered inevitable only depending on a 5-year of adjuvant endocrine therapy. Therefore, extended endocrine therapy is considered as a possible measure to reduce the risk of recurrence.

Numerous clinical studies have focused on extended endocrine therapy in patients with specific types of breast cancer. In 2017, the National Comprehensive Cancer Network (NCCN) updated the recommends for extended endocrine therapy with aromatase inhibitor, where postmenopausal early-stage breast cancer patients wo have high risk factors may be considered to be given an extended 5-year endocrine treatment with aromatase inhibitor after the initial 5-year treatment. In 2019, the Chinese Society of Clinical Oncology also suggested that postmenopausal hormone receptor-positive patients who have been well tolerated to the initial 5 years of adjuvant endocrine therapy can be given the extended endocrine therapy under some restrictions.

However, extended endocrine therapy may also cause other risks in patients. Long-term tamoxifen treatment can significantly increase the incidence of adverse reactions such as endometrial cancer, thrombotic disease, and dyslipidemia, and long-term aromatase inhibitor treatment can also increase the incidence of osteoporosis, fractures, dyslipidemia, and hypertension. Although anti-cancer treatment can reduce cancer deaths, it may increase deaths due to cardiovascular diseases.

An attempt has been proposed to find out an indicator that can effectively determine the necessity of extended endocrine therapy in such patients, not only improving the prognosis of breast cancer patients, but also reducing treatment-related side effects. The author's team recently discovered sj-subway, a possible factor with a long tubular structure in breast cancer lesions. The authors found that the higher expression of sj-subway indicates the worse patient's prognosis. So the positive expression of sj-subway may be a predictor of recurrence and metastasis in high-risk hormone receptor-positive patients. However, whether this predictor can be used clinically remains to be studied.

This real-world study intends to analyze the difference in the clinical efficacy of extended endocrine therapy under different sj-subway expression in high-risk hormone receptor-positive breast cancer patients, and to explore whether sj-subway can screen out the patients who can benefit from extended endocrine therapy, thus providing a therapeutic help for hormone receptor-positive breast cancer patients.

DETAILED DESCRIPTION:
Breast cancer has been one of the most common malignant tumors in women, accounting for 23% of all the malignancies. There are estimated 1,300,000 new cases of breast cancers and 400,000 deaths due to breast cancers every year in the world. Hormone receptor-positive breast cancer accounts for about 70% of all breast cancers.

Since ovarian resection was first used in the treatment of advanced breast cancer in the late 19th century, with more than a century of development, endocrine therapy has become the most important adjuvant therapy for hormone receptor-positive breast cancers, especially for advanced breast cancers. Increasing clinical trials of adjuvant endocrine therapy such as ATAC, BIG1-98, and IES, which have been implemented since 2002, have ascertained the effect of adjuvant endocrine therapy with aromatase inhibitor, and the guidelines for the diagnosis and treatment of breast cancer have been also changed accordingly.

Although early-stage hormone receptor-positive breast cancer patients have a better prognosis than HER-2 positive and triple-negative patients, there is still a long-lasting risk of postoperative recurrence, which has been confirmed in two large-scale meta-analyses reported by the Early Breast Cancer Trialists' Collaborative Group (EBCTCG). A meta-analysis released by the EBCTCG in 1998 indicated that early-stage hormone receptor-positive breast cancer patients, especially lymph node-positive patients, experienced the second recurrence peak at 2-3 years and 7-9 years after completion of endocrine therapy. In 2016, the EBCTCG released another relevant study at the annual meeting of the American Society of Clinical Oncology (ASCO), in which the long-term recurrence rate within 5-20 years was up to 14% in T1N0 breast cancer patients who had undergone 5 years of adjuvant endocrine therapy. Therefore, the 5 years of standard adjuvant endocrine therapy cannot eliminate the risk of recurrence. Most scholars have suggested that the duration of endocrine therapy should be extended to reduce the recurrence risk of breast cancer.

Numerous clinical trials have focused on the use of extended endocrine therapy in patients with specific types of breast cancer. In the MA17R trial, patients received 3-5 years of tamoxifen or 5 years of aromatase inhibitor treatment, followed by another 5 years of aromatase inhibitor treatment. The extended aromatase inhibitor treatment was found to significantly improve the disease-free survival time of hormone receptor-positive early breast cancer patients, while also reducing the risk of contralateral breast cancer and distant relapse. In the NSABP B42 trial, patients who had received initial 5 years of aromatase inhibitor treatment or initial 5 years of tamoxifen + aromatase inhibitor treatment were all treated with extended aromatase inhibitor. Although the primary endpoint (P = 0.048) did not reach the expected value, extended treatment with aromatase inhibitors significantly reduced the secondary endpoints - breast cancer-free interval and distant relapse, confirming the conclusion of the MA17R study. In the DATA trial, although extended treatment with aromatase inhibitor did not benefit in general, subgroup analysis showed that some high-risk patients, such as patients with positive lymph nodes, tumors larger than 2 cm in diameter, or receiving chemotherapy, could benefit from 6 years of anastrozole treatment. The IDEAL trial showed that there is a trend of benefit in patients with positive lymph nodes. With the support of many large-scale clinical studies published in succession, the NCCN practice guidelines for breast cancer released in 2017 recommends an additional 5 years of aromatase inhibitor treatment following the initial 5-year treatment in postmenopausal patients with early-stage breast cancer at high risk for relapse. As per the Chinese Society of Clinical Oncology guidelines published in 2019, the extended endocrine therapy is also recommended for postmenopausal hormone receptor-positive patients who have been well tolerated to the initial 5-year adjuvant treatment. However, there are some restrictions, such as positive lymph nodes, G3 or other risk factors that require adjuvant chemotherapy. For premenopausal hormone receptor-positive patients who have been well tolerated to the initial 5 years of endocrine treatment, extended endocrine therapy is also recommended in some situations, such as the presence of positive lymph nodes, G3, less than 35 years old at diagnosis, high-level Ki-67 or pT2 and above.

However, the extended endocrine therapy also has some adverse events. Multiple studies have shown that long-term use of tamoxifen can significantly increase the incidence of adverse reactions such as endometrial cancer, thrombotic disease, and dyslipidemia. Similarly, long-term treatment with aromatase inhibitors can also increase the incidence of adverse reactions such as osteoporosis, fractures, dyslipidemia, and hypertension. In the ATLAS trial, the incidence of endometrial cancer in patients treated with 10 years of tamoxifen was higher than that in patients treated with 5 years of tamoxifen. Similar results are discovered in the aTTom trial. In the IDEAL trial, the incidence rates of osteoarthritis and osteoporosis in patients treated with 5 years of letrozole was increased by 14% and 10% of that in patients undergoing 2.5 years of treatment. A study involving nearly 100,000 breast cancer patients showed that only 49.9% of breast cancer patients died of breast cancer, 16.3% died of cardiovascular disease, and 33.8% died of other causes. Among them, breast cancer and cardiovascular disease were the main causes of death in well- and poor-tolerated patients, respectively. This suggests that although anti-cancer treatment can reduce cancer deaths, it may increase the death due to cardiovascular disease. Such deaths are often offset, which often improves the BCFI, but does not benefit the overall survival.

Therefore, an effective predictor for relapse risks that can accurately determine the necessity of extended endocrine therapy is expected to be discovered. The use of this predictor will both improve patient's prognosis and reduce treatment-related side effects. The author's team recently discovered a possible factor with a long tubular structure in breast cancer lesions using immunofluorescence staining, which was named as sj-subway. The authors conducted a retrospective analysis based on the specimen library and case follow-up library of the Breast Center of Shengjing Hospital Affiliated to China Medical University. They found that sj-subway was positively expressed in various subtypes of breast cancer tissues, and mostly expressed in the hormone receptor-positive subtype. The group with more sj-subway expression had a higher positive expression of hormone receptor/ progesterone receptor. Further survival analysis also revealed the worse prognosis of patients with the existence of higher sj-subway expression. Therefore, the authors speculate that positively expressed sj-subway may become a predictor of recurrence and metastasis in high-risk patients with hormone receptor positive. However, the clinical use of this factor to screen the population benefiting from extended endocrine therapy remains to be studied.

This real-world study intends to observe the difference in the clinical efficacy of extended endocrine therapy under different sj-subway expression in high-risk hormone receptor-positive breast cancer patients, and to analyze whether the use of sj-subway can further screen out the population with benefit from extended endocrine therapy, thus further improving the survival of such patients without additional adverse events.

ELIGIBILITY:
Inclusion Criteria:

* early-stage invasive breast cancer positive for estrogen receptor and / or progesterone receptor is pathologically confirmed;
* patients who have completed standard endocrine therapy for 5 years without recurrence and metastasis;
* 18-70 years old;
* patients with one of the following six manifestations: KI67 ≥ 30%; tumor size > 2 cm; positive lymph nodes; histological grade III; vascular cancer thrombus; HER-2 gene overexpression or amplification.

Exclusion Criteria:

* with a history of other malignancies;
* patients who have severe abnormalities in important organs, such as the heart, liver, and kidney or who cannot be tolerant to extended treatment due to poor constitution;
* patients with severe osteoporosis or dyslipidemia, or those who cannot tolerate endocrine therapy ;
* patients who have participated in other clinical trials.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The early-stage invasive breast cancer positive for estrogen receptor and / or progesterone receptor and have completed standard endocrine therapy for 5 years.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-07-19 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 5 years after enrollment
  the time from enrollment to relapse or death due to any reason.

SECONDARY OUTCOMES:
Overall survival | 5 years after enrollment
  the time from enrollment to death due to any reason
Incidence of contralateral breast cancer | 1, 2, 3, 4, and 5 years after enrollment
  the proportion of contralateral breast cancer. Evaluations will be made at 1, 2, 3, 4, and 5 years after enrollment
Incidence of adverse events | 1, 2, 3, 4, and 5 years after enrollment
  the proportion of adverse events, including osteoporosis, bone pain, fractures, dyslipidemia, endometrial lesions. Evaluations will be made 1, 2, 3, 4, and 5 years after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Qi Xue, Principal Investigator — Shengjing Hospital; Xi Gu, Principal Investigator — Shengjing Hospital; Nan Niu, Principal Investigator — Shengjing Hospital; Tian-Hui Xia, Principal Investigator — Shengjing Hospital; Wei Tu, Principal Investigator — Fourth Affiliated Hospital of China Medical University; Hong Xu, Principal Investigator — Liaoning Cancer Hospital & Institute; Hao Zhang, Principal Investigator — Liaoning Cancer Hospital & Institute; Yuan-Xi Huang, Principal Investigator — Heilongjiang Cancer Hospital; Shao-Qiang Cheng, Principal Investigator — Heilongjiang Cancer Hospital; Bing-Shu Xia, Principal Investigator — Heilongjiang Cancer Hospital; Wen-Bin Guo, Principal Investigator — Dalian Municipal Central Hospital; Xue Jiang, Principal Investigator — Dalian Municipal Central Hospital
Locations (10):
- China (10):
  - Cancer Hospital Affiliated to Harbin Medical University, Harbin, Heilongjiang
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - Panjin Liaohe Oilfield Gem Flower Hospital, Panjin, Liaoning
  - Shengjing Hospital affiliated to China Medical University, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Liaoning Tumor Hospital & Institute, Shenyang, Liaoning
  - People's Hospital of Liaoning Province, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: Undecided